CLINICAL TRIAL: NCT03449953
Title: Critical Care Outcomes of Patients With Hematologic Malignancy and Hematopoietic Cell Transplantation
Brief Title: Critical Care Outcomes of Hematologic Oncology Patients
Acronym: COHO
Status: Active, not recruiting | Type: Observational
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: COHO vOct2017
Record Dates: First submitted 2017-11-23; First posted 2018-02-28 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Hematologic Malignancy; Stem Cell Transplant
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hematologic malignancy patients are admitted to ICU in increasing numbers. Successful ICU intervention has led to an increasing number of ICU survivors; however, there is a lack of information available about these patients' long term survival and quality of life. There is little Canadian data regarding ICU survival and regarding 1-year survival and functional outcomes in this group of patients. Over 500 patients are admitted annually to Canadian ICUs with an underlying hematologic malignancy or stem cell transplant, yet there is a paucity of up to date long-term outcome data. This information will facilitate a better understanding who would best benefit from critical care interventions and the impact of critical illness on their level of function at 1 year as well as survival.

DETAILED DESCRIPTION:
At the time of ICU admission, the investigators will collect clinical data from the medical chart on a daily basis including demographics, pre-existing disease(s), treatment and reason for ICU admission.

At the time of ICU discharge, the investigators will measure exercise tolerance and quality of life at 3 time intervals (Phase 2).

For Phase 2, patients will be seen at day 7 following ICU discharge, 6 months following ICU discharge and 12 months after ICU discharge during their routine oncology follow up visits. During these visits, they will undergo a functional assessment (6 minute walk test) and questionnaires to determine their quality of life following ICU (validated outcome measures).

All patients will complete outcome measures 1 to 5 below; Outcome measures 1 to 3 will be administered at 7 days and 1 to 5 at 6 months and 12 months after ICU discharge.

Validated Outcomes Measures:

1. Functional Independence Measure (FIM): a patient-centered measure of functional disability that captures burden of care on a daily basis and involves motor (FIM-motor) and cognitive function (FIM-cognition). FIM predicts disability outcome and rehabilitation needs in diverse patient populations.
2. Six Minute Walk Test (6MWT) with continuous oximetry to measure the oxygen saturation of arterial blood will be performed to assess exercise capacity. It is simple to execute, inexpensive, standardized and gives a tangible measure of functional exercise capacity because it uses an exercise mode that is relevant to everyday activities.
3. Clinical Frailty Scale (CFS): CFS is a 9-category tool ranging from 1 (Very fit) to 9 (Terminally ill). It provides predictive information about death or need for an institution. It is easy to administer in less than 5 minutes.
4. Medical Outcomes Study Short Form - 36 Questionnaire (SF-36): SF-36 evaluates 8 health concepts: physical functioning, role functioning-physical, bodily pain, general health, vitality, social functioning, role functioning- emotional, mental health and reported health transition. It has been validated in diverse patient populations and is a responsive and reproducible instrument; and can be completed in less than 15 minutes.
5. FACT-BMT: A 47-item, valid and reliable measure of five dimensions of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >16 years with Hematologic Malignancy (HM) or post Stem Cell Transplant (HCT) who require ICU admission.
* HM includes: acute myeloid leukemia, acute lymphocytic leukemia, chronic myeloid leukemia, chronic lymphocytic leukemia, myeloma, lymphoma, myelofibrosis, and other myeloproliferative disorders or myelodysplastic syndromes.
* HCT is defined as the transplantation of multipotent hematopoietic stem cells from bone marrow, peripheral blood, or umbilical cord blood.

Exclusion Criteria:

* Subjects with significant preexisting neurological or psychiatric disease will be excluded from Phase 2 (1-year follow-up) but will be included in Phase 1.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematologic malignancy (HM) and hematopoietic cell transplantation (HCT) frequently develop life-threatening illness and require admission to an intensive care unit (ICU). In light of advancements in care and extension of treatments to much higher risk candidates, survival and functional outcome evaluation become crucial for informed development of practice guidelines to guide pre-ICU risk stratification, as well as ICU and post-ICU care. Robust and up to date long-term data on ICU morbidity and mortality outcomes are lacking.
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
1 year survival | 1 year
  1 year survival in enrolled patients

SECONDARY OUTCOMES:
Intensive Care Unit survival | 1 year
  ICU survival in enrolled patients
6 month functional outcome measured by the 6 minute walk test (6MWT) | 6 months
  6MWT will be performed to assess exercise capacity at 6 months
6 month Functional Independent Measure questionnaire (FIM) | 6 months
  FIM: Captures burden of care on a daily basis and involves motor and cognitive function. FIM predicts disability outcome and rehabilitation needs.
6 month Clinical Frailty Scale (CFS) | 6 months
  CFS: Is a 9-category tool ranging from 1 (Very fit) to 9 (Terminally ill). It provides predictive information about death or need for an institution
6 month Short Form 36 Health Questionnaire (SF 36) | 6 months
  SF-36: Evaluates 8 health concepts: physical functioning, role functioning-physical, bodily pain, general health, vitality, social functioning, role functioning- emotional, mental health and reported health transition.
6 month Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT BMT) | 6 months
  FACT-BMT: A 47-item, valid and reliable measure of five dimensions of quality of life.
1 year functional outcome measured by the 6 minute walk test (6MWT) | 1 year
  6MWT will be performed to assess exercise capacity at 6 months
1 year Functional Independent Measure questionnaire (FIM) | 1 year
  FIM: Captures burden of care on a daily basis and involves motor and cognitive function. FIM predicts disability outcome and rehabilitation needs.
1 year Clinical Frailty Scale (CFS) | 1 year
  CFS: Is a 9-category tool ranging from 1 (Very fit) to 9 (Terminally ill). It provides predictive information about death or need for an institution
1 year Short Form 36 Health Questionnaire (SF 36) | 1 year
  SF-36: Evaluates 8 health concepts: physical functioning, role functioning-physical, bodily pain, general health, vitality, social functioning, role functioning- emotional, mental health and reported health transition.
1 year Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT BMT) | 1 year
  FACT-BMT: A 47-item, valid and reliable measure of five dimensions of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Laveena Munshi, MD, FRCPC, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (13):
- Canada (13):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guidelines for intensive care unit admission, discharge, and triage. Task Force of the American College of Critical Care Medicine, Society of Critical Care Medicine. Crit Care Med. 1999 Mar;27(3):633-8. PMID 10199547
- [Background] Roze des Ordons AL, Chan K, Mirza I, Townsend DR, Bagshaw SM. Clinical characteristics and outcomes of patients with acute myelogenous leukemia admitted to intensive care: a case-control study. BMC Cancer. 2010 Sep 28;10:516. doi: 10.1186/1471-2407-10-516. PMID 20920175
- [Background] Cornish M, Butler MB, Green RS. Predictors of Poor Outcomes in Critically Ill Adults with Hematologic Malignancy. Can Respir J. 2016;2016:9431385. doi: 10.1155/2016/9431385. Epub 2016 Feb 24. PMID 27445571
- [Background] Kraguljac AP, Croucher D, Christian M, Ibrahimova N, Kumar V, Jacob G, Kiss A, Minden MD, Mehta S. Outcomes and Predictors of Mortality for Patients with Acute Leukemia Admitted to the Intensive Care Unit. Can Respir J. 2016;2016:3027656. doi: 10.1155/2016/3027656. Epub 2016 Jun 30. PMID 27445524
- [Background] Trinkaus MA, Lapinsky SE, Crump M, Keating A, Reece DE, Chen C, Hallett DC, Franke N, Winter A, Mikhael JR. Predictors of mortality in patients undergoing autologous hematopoietic cell transplantation admitted to the intensive care unit. Bone Marrow Transplant. 2009 Mar;43(5):411-5. doi: 10.1038/bmt.2008.336. Epub 2008 Oct 20. PMID 18936734
- [Background] Scales DC, Thiruchelvam D, Kiss A, Sibbald WJ, Redelmeier DA. Intensive care outcomes in bone marrow transplant recipients: a population-based cohort analysis. Crit Care. 2008;12(3):R77. doi: 10.1186/cc6923. Epub 2008 Jun 11. PMID 18547422
- [Background] Yadav H, Nolan ME, Bohman JK, Cartin-Ceba R, Peters SG, Hogan WJ, Gajic O, Kor DJ. Epidemiology of Acute Respiratory Distress Syndrome Following Hematopoietic Stem Cell Transplantation. Crit Care Med. 2016 Jun;44(6):1082-90. doi: 10.1097/CCM.0000000000001617. PMID 26807683
- [Background] Thakkar SG, Fu AZ, Sweetenham JW, Mciver ZA, Mohan SR, Ramsingh G, Advani AS, Sobecks R, Rybicki L, Kalaycio M, Sekeres MA. Survival and predictors of outcome in patients with acute leukemia admitted to the intensive care unit. Cancer. 2008 May 15;112(10):2233-40. doi: 10.1002/cncr.23394. PMID 18348307
- [Background] Cuthbertson BH, Rajalingam Y, Harrison S, McKirdy F, On behalf of the Scottish Intensive Care Society. The outcome of haematological malignancy in Scottish intensive care units. JICS 2008; 9 (2)
- [Background] Bird GT, Farquhar-Smith P, Wigmore T, Potter M, Gruber PC. Outcomes and prognostic factors in patients with haematological malignancy admitted to a specialist cancer intensive care unit: a 5 yr study. Br J Anaesth. 2012 Mar;108(3):452-9. doi: 10.1093/bja/aer449. Epub 2012 Jan 31. PMID 22298243
- [Background] Hampshire PA, Pugh R, Hajimichael P. Outcomes for critically ill patients with haematological malignancies in specialist and non-specialist centres in the United Kingdom. Journal of Cancer Therapeutics & Research 2014, http://www.hoajonline.com/journals/pdf/2049-7962-3-5.pdf
- [Background] Grgic Medic M, Gornik I, Gasparovic V. Hematologic malignancies in the medical intensive care unit--Outcomes and prognostic factors. Hematology. 2015 Jun;20(5):247-53. doi: 10.1179/1607845414Y.0000000206. Epub 2014 Oct 13. PMID 25310461
- [Background] Azoulay E, Mokart D, Pene F, Lambert J, Kouatchet A, Mayaux J, Vincent F, Nyunga M, Bruneel F, Laisne LM, Rabbat A, Lebert C, Perez P, Chaize M, Renault A, Meert AP, Benoit D, Hamidfar R, Jourdain M, Darmon M, Schlemmer B, Chevret S, Lemiale V. Outcomes of critically ill patients with hematologic malignancies: prospective multicenter data from France and Belgium--a groupe de recherche respiratoire en reanimation onco-hematologique study. J Clin Oncol. 2013 Aug 1;31(22):2810-8. doi: 10.1200/JCO.2012.47.2365. Epub 2013 Jun 10. PMID 23752112
- [Background] Mokart D, Darmon M, Resche-Rigon M, Lemiale V, Pene F, Mayaux J, Rabbat A, Kouatchet A, Vincent F, Nyunga M, Bruneel F, Lebert C, Perez P, Renault A, Hamidfar R, Jourdain M, Meert AP, Benoit D, Chevret S, Azoulay E. Prognosis of neutropenic patients admitted to the intensive care unit. Intensive Care Med. 2015 Feb;41(2):296-303. doi: 10.1007/s00134-014-3615-y. Epub 2015 Jan 13. PMID 25578678
- [Background] Lengline E, Chevret S, Moreau AS, Pene F, Blot F, Bourhis JH, Buzyn A, Schlemmer B, Socie G, Azoulay E. Changes in intensive care for allogeneic hematopoietic stem cell transplant recipients. Bone Marrow Transplant. 2015 Jun;50(6):840-5. doi: 10.1038/bmt.2015.55. Epub 2015 Mar 23. PMID 25798675
- [Background] Lemiale V, Resche-Rigon M, Mokart D, Pene F, Rabbat A, Kouatchet A, Vincent F, Bruneel F, Nyunga M, Lebert C, Perez P, Meert AP, Benoit D, Chevret S, Azoulay E. Acute respiratory failure in patients with hematological malignancies: outcomes according to initial ventilation strategy. A groupe de recherche respiratoire en reanimation onco-hematologique (Grrr-OH) study. Ann Intensive Care. 2015 Dec;5(1):28. doi: 10.1186/s13613-015-0070-z. Epub 2015 Sep 30. PMID 26429355
- [Background] Champigneulle B, Merceron S, Lemiale V, Geri G, Mokart D, Bruneel F, Vincent F, Perez P, Mayaux J, Cariou A, Azoulay E. What is the outcome of cancer patients admitted to the ICU after cardiac arrest? Results from a multicenter study. Resuscitation. 2015 Jul;92:38-44. doi: 10.1016/j.resuscitation.2015.04.011. Epub 2015 Apr 24. PMID 25917260
- [Background] Herridge MS, Chu LM, Matte A, Tomlinson G, Chan L, Thomas C, Friedrich JO, Mehta S, Lamontagne F, Levasseur M, Ferguson ND, Adhikari NK, Rudkowski JC, Meggison H, Skrobik Y, Flannery J, Bayley M, Batt J, Santos CD, Abbey SE, Tan A, Lo V, Mathur S, Parotto M, Morris D, Flockhart L, Fan E, Lee CM, Wilcox ME, Ayas N, Choong K, Fowler R, Scales DC, Sinuff T, Cuthbertson BH, Rose L, Robles P, Burns S, Cypel M, Singer L, Chaparro C, Chow CW, Keshavjee S, Brochard L, Hebert P, Slutsky AS, Marshall JC, Cook D, Cameron JI; RECOVER Program Investigators (Phase 1: towards RECOVER); Canadian Critical Care Trials Group. The RECOVER Program: Disability Risk Groups and 1-Year Outcome after 7 or More Days of Mechanical Ventilation. Am J Respir Crit Care Med. 2016 Oct 1;194(7):831-844. doi: 10.1164/rccm.201512-2343OC. PMID 26974173
- [Background] Heyland DK, Garland A, Bagshaw SM, Cook D, Rockwood K, Stelfox HT, Dodek P, Fowler RA, Turgeon AF, Burns K, Muscedere J, Kutsogiannis J, Albert M, Mehta S, Jiang X, Day AG. Recovery after critical illness in patients aged 80 years or older: a multi-center prospective observational cohort study. Intensive Care Med. 2015 Nov;41(11):1911-20. doi: 10.1007/s00134-015-4028-2. Epub 2015 Aug 26. PMID 26306719
- [Background] Bekelman JE, Halpern SD, Blankart CR, Bynum JP, Cohen J, Fowler R, Kaasa S, Kwietniewski L, Melberg HO, Onwuteaka-Philipsen B, Oosterveld-Vlug M, Pring A, Schreyogg J, Ulrich CM, Verne J, Wunsch H, Emanuel EJ; International Consortium for End-of-Life Research (ICELR). Comparison of Site of Death, Health Care Utilization, and Hospital Expenditures for Patients Dying With Cancer in 7 Developed Countries. JAMA. 2016 Jan 19;315(3):272-83. doi: 10.1001/jama.2015.18603. PMID 26784775
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Wise MP, Barnes RA, Baudouin SV, Howell D, Lyttelton M, Marks DI, Morris EC, Parry-Jones N; British Committee for Standards in Haematology. Guidelines on the management and admission to intensive care of critically ill adult patients with haematological malignancy in the UK. Br J Haematol. 2015 Oct;171(2):179-188. doi: 10.1111/bjh.13594. Epub 2015 Aug 19. No abstract available. PMID 26287443
- [Background] Mehta S, Burry L, Cook D, Fergusson D, Steinberg M, Granton J, Herridge M, Ferguson N, Devlin J, Tanios M, Dodek P, Fowler R, Burns K, Jacka M, Olafson K, Skrobik Y, Hebert P, Sabri E, Meade M; SLEAP Investigators; Canadian Critical Care Trials Group. Daily sedation interruption in mechanically ventilated critically ill patients cared for with a sedation protocol: a randomized controlled trial. JAMA. 2012 Nov 21;308(19):1985-92. doi: 10.1001/jama.2012.13872. PMID 23180503
- [Background] Liu J, Bell C, Campbell V, DeBacker J, Tamberg E, Lee C, Mehta S. Noninvasive Ventilation in Patients With Hematologic Malignancy. J Intensive Care Med. 2017 Jan 1:885066617690725. doi: 10.1177/0885066617690725. Online ahead of print. PMID 28142306
- [Background] MacEachern KN, Kraguljac AP, Mehta S. Nutrition Care of Critically Ill Patients with Leukemia: A Retrospective Study. Can J Diet Pract Res. 2019 Mar 1;80(1):34-38. doi: 10.3148/cjdpr-2018-033. Epub 2018 Nov 15. PMID 30430851
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Oczkowski WJ, Barreca S. The functional independence measure: its use to identify rehabilitation needs in stroke survivors. Arch Phys Med Rehabil. 1993 Dec;74(12):1291-4. doi: 10.1016/0003-9993(93)90081-k. PMID 8259894
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Ware JE J, Kosinski M, Gandek B. SF-36 Health Survey: manual and interpretation guide. Lincoln,R.I.: QualityMetric Inc.; 2002.
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] McQuellon RP, Russell GB, Cella DF, Craven BL, Brady M, Bonomi A, Hurd DD. Quality of life measurement in bone marrow transplantation: development of the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) scale. Bone Marrow Transplant. 1997 Feb;19(4):357-68. doi: 10.1038/sj.bmt.1700672. PMID 9051246
- [Background] Brazier J, Roberts J, Deverill M. The estimation of a preference-based measure of health from the SF-36. J Health Econ. 2002 Mar;21(2):271-92. doi: 10.1016/s0167-6296(01)00130-8. PMID 11939242
- [Background] Ferguson ND, Scales DC, Pinto R, Wilcox ME, Cook DJ, Guyatt GH, Schunemann HJ, Marshall JC, Herridge MS, Meade MO; Canadian Critical Care Trials Group. Integrating mortality and morbidity outcomes: using quality-adjusted life years in critical care trials. Am J Respir Crit Care Med. 2013 Feb 1;187(3):256-61. doi: 10.1164/rccm.201206-1057OC. Epub 2012 Nov 29. PMID 23204250
- [Background] Bender JM, Ampofo K, Gesteland P, Stoddard GJ, Nelson D, Byington CL, Pavia AT, Srivastava R. Development and validation of a risk score for predicting hospitalization in children with influenza virus infection. Pediatr Emerg Care. 2009 Jun;25(6):369-75. doi: 10.1097/PEC.0b013e3181a792a9. PMID 19458562
- [Background] Sullivan LM, Massaro JM, D'Agostino RB Sr. Presentation of multivariate data for clinical use: The Framingham Study risk score functions. Stat Med. 2004 May 30;23(10):1631-60. doi: 10.1002/sim.1742. PMID 15122742
- [Background] Hanley JA, McNeil BJ. A method of comparing the areas under receiver operating characteristic curves derived from the same cases. Radiology. 1983 Sep;148(3):839-43. doi: 10.1148/radiology.148.3.6878708.
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008